CLINICAL TRIAL: NCT03976401
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Efruxifermin in Subjects With Nonalcoholic Steatohepatitis (NASH)
Brief Title: A Study of Efruxifermin in Subjects With Histologically Confirmed Nonalcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akero Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK-US-001-0101
Record Dates: First submitted 2019-06-03; First posted 2019-06-06 (Actual); Results first posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- EFX Dose 1 (Experimental): Main Study
  Interventions: Drug: EFX
- EFX Dose 2 (Experimental): Main Study
  Interventions: Drug: EFX
- EFX Dose 3 (Experimental): Main Study
  Interventions: Drug: EFX
- Placebo (Placebo Comparator): Main Study
  Interventions: Drug: Placebo
- EFX Dose (Cohort C) (Experimental)
  Interventions: Drug: EFX
- Placebo (Cohort C) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EFX — Administered by subcutaneous injection
  Arms: EFX Dose (Cohort C); EFX Dose 1; EFX Dose 2; EFX Dose 3
Drug: Placebo — Administered by subcutaneous injection
  Arms: Placebo; Placebo (Cohort C)

SUMMARY:
This is a multi-center evaluation of efruxifermin (EFX) in a randomized, double-blind, placebo-controlled study administered for 16 weeks in subjects with biopsy proven F1 - F4 NASH.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and non-pregnant, non-lactating females between 18 - 80 years of age inclusive, based on the date of the screening visit.
* Main Study only: Body mass index (BMI) > 25 kg/m^2 (unless the patient has biopsy-proven NASH documented within the last 2 years).
* Main Study only: Must have confirmation of ≥ 10% liver fat content on magnetic resonance imaging- proton density fat fraction (MRI-PDFF) at screening.
* Main Study only: Biopsy-proven NASH. Must have had a liver biopsy within 180 days of randomization with fibrosis stage 1 to 3 and a non-alcoholic fatty liver disease (NAFLD) activity score (NAS) of ≥ 4 with at least a score of 1 in each of the following NAS components:

  * Steatosis (scored 0 to 3),
  * Ballooning degeneration (scored 0 to 2), and
  * Lobular inflammation (scored 0 to 3)
* Cohort C only: FibroScan® measurement > 13.1 kPa.
* Cohort C only: Cirrhosis due to NASH. Liver biopsy consistent with F4 fibrosis according to the NAS system, confirmed by the central or local reader.

Exclusion Criteria:

* Weight gain or loss > 5% in the 3 months prior to randomization or > 10% in the 6 months prior to screening.
* Type 1 and insulin-dependent Type 2 diabetes.
* Poorly controlled hypertension (blood pressure > 160/100).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2022-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (24):
  - Akero Clinical Study Site, Tucson, Arizona
  - Akero Clinical Study Site, Little Rock, Arkansas
  - Akero Clinical Study Site, Huntington Park, California
  - Akero Clinical Study Site, Los Angeles, California
  - Akero Clinical Study Site, Panorama City, California
  - Akero Clinical Study Site, Poway, California
  - Akero Clinical Study Site, Boca Raton, Florida
  - Akero Clinical Study Site, Lakewood Rch, Florida
  - Akero Clinical Study Site, Miami, Florida
  - Akero Clinical Study Site, New Port Richey, Florida
  - Akero Clinical Study Site, Ocoee, Florida
  - Akero Clinical Study Site, Port Orange, Florida
  - Akero Clinical Study Site, Sarasota, Florida
  - Akero Clinical Study Site, Baton Rouge, Louisiana
  - Akero Clinical Study Site, Marrero, Louisiana
  - Akero Clinical Study Site, Kansas City, Missouri
  - Akero Clinical Study Site, Berlin, New Jersey
  - Akero Clinical Study Site, Chattanooga, Tennessee
  - Akero Clinical Study Site, Cedar Park, Texas
  - Akero Clinical Study Site, Dallas, Texas
  - Akero Clinical Study Site, Edinburg, Texas
  - Akero Clinical Study Site, Fort Worth, Texas
  - Akero Clinical Study Site, San Antonio, Texas
  - Akero Clinical Study Site, Webster, Texas
- Akero Clinical Study Site, San Juan, Puerto Rico

REFERENCES:
- [Derived] Alkhouri N, Beyer C, Shumbayawonda E, Andersson A, Yale K, Rolph T, Chung RT, Vuppalanchi R, Cusi K, Loomba R, Pansini M, Dennis A. Decreases in cT1 and liver fat content reflect treatment-induced histological improvements in MASH. J Hepatol. 2025 Mar;82(3):438-445. doi: 10.1016/j.jhep.2024.08.031. Epub 2024 Sep 25. PMID 39326675
- [Derived] Harrison SA, Ruane PJ, Freilich B, Neff G, Patil R, Behling C, Hu C, Shringarpure R, de Temple B, Fong E, Tillman EJ, Rolph T, Cheng A, Yale K. A randomized, double-blind, placebo-controlled phase IIa trial of efruxifermin for patients with compensated NASH cirrhosis. JHEP Rep. 2022 Aug 23;5(1):100563. doi: 10.1016/j.jhepr.2022.100563. eCollection 2023 Jan. PMID 36644237
- [Derived] Harrison SA, Ruane PJ, Freilich BL, Neff G, Patil R, Behling CA, Hu C, Fong E, de Temple B, Tillman EJ, Rolph TP, Cheng A, Yale K. Efruxifermin in non-alcoholic steatohepatitis: a randomized, double-blind, placebo-controlled, phase 2a trial. Nat Med. 2021 Jul;27(7):1262-1271. doi: 10.1038/s41591-021-01425-3. Epub 2021 Jul 8. PMID 34239138

RESULTS

PARTICIPANT FLOW:
Groups:
- Main Study EFX 28 mg; Main Study EFX 50 mg; Main Study EFX 70 mg; Main Study Placebo; Cohort C EFX 50 mg; Cohort C Placebo: QW SC injection for 16 weeks.
Period: Overall Study
Arm/Group | Main Study EFX 28 mg | Main Study EFX 50 mg | Main Study EFX 70 mg | Main Study Placebo | Cohort C EFX 50 mg | Cohort C Placebo
Started | 19 | 20 | 20 | 21 | 20 | 10
Completed | 16 | 16 | 15 | 19 | 19 | 9
Not Completed | 3 | 4 | 5 | 2 | 1 | 1
Not completed — Adverse Event | 2 | 0 | 4 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (All randomized subjects)
Groups:
- Main EFX 28 mg; Main EFX 50 mg; Main EFX 70 mg: Main Study
  EFX: Administered by subcutaneous injection
- Main Placebo: Main Study
  Placebo: Administered by subcutaneous injection
- Cohort C EFX 50 mg: Cohort C
  EFX: Administered by subcutaneous injection
- Cohort C Placebo: Cohort C
  Placebo: Administered by subcutaneous injection
- Total: Total of all reporting groups
Arm/Group | Main EFX 28 mg | Main EFX 50 mg | Main EFX 70 mg | Main Placebo | Cohort C EFX 50 mg | Cohort C Placebo | Total
Number analyzed (Participants) | 19 | 20 | 20 | 21 | 20 | 10 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (12.40) | 52.6 (14.19) | 53.0 (13.22) | 52.4 (9.57) | 61.1 (10.0) | 57.1 (14.4) | 54.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 11 | 15 | 16 | 3 | 65
  Male | 9 | 10 | 9 | 6 | 4 | 7 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 7 | 10 | 8 | 5 | 53
  Not Hispanic or Latino | 7 | 9 | 13 | 11 | 12 | 5 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 2 | 1 | 1 | 1 | 0 | 5
  White | 19 | 18 | 19 | 19 | 18 | 10 | 103
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 20 | 21 | 20 | 10 | 110

OUTCOME MEASURES:

1. Primary Outcome: Main: Absolute Change From Baseline in Hepatic Fat Fraction Assessed by MRI-PDFF at Week 12.
Description: Main study. ANCOVA multiple imputation with treatment group and F1 fibrosis score (F1 vs F2-3) as factors and baseline hepatic fat fraction measured by MRI-PDFF as a covariate.
Time Frame: 12 weeks
Population: Full Analysis Set (all randomized subjects)
Measure: Least Squares Mean (Standard Error); unit: Absolute percentage of hepatic fat
Arm/Group | Main Study EFX 28 mg | Main Study EFX 50 mg | Main Study EFX 70 mg | Main Study Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Absolute percentage of hepatic fat | -12.32 (1.04) | -13.44 (1.04) | -14.14 (1.04) | -0.29 (0.98)

2. Secondary Outcome: Main: Absolute Change From Baseline in Hepatic Fat Fraction Assessed by MRI-PDFF at Week 22-24.
Description: Main study. Included subjects with ≥30% relative fat reduction on MRI-PDFF at Week 12 that were required to return between Weeks 22 - 24. ANCOVA model with treatment group and F1 fibrosis score (F1 vs F2-3) as factors and baseline hepatic fat fraction as a covariate were performed.
Time Frame: 22-24 weeks
Population: Subjects from Full Analysis Set with 30% or greater reduction in hepatic fat fraction at Week 12, who returned for MRI-PDFF
Measure: Least Squares Mean (Standard Error); unit: Absolute percentage of hepatic fat
Arm/Group | Main Study EFX 28 mg | Main Study EFX 50 mg | Main Study EFX 70 mg | Main Study Placebo
Number analyzed (Participants) | 16 | 17 | 15 | 2
Absolute percentage of hepatic fat | -9.50 (1.49) | -8.99 (1.49) | -12.72 (1.50) | -14.45 (4.08)

3. Secondary Outcome: Main: Percent Change From Baseline in Hepatic Fat Fraction Measured by MRI-PDFF at Week 12.
Description: as for outcome 1
Time Frame: 12 weeks
Population: Full Analysis Set (all randomized subjects)
Measure: Least Squares Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Main Study EFX 28 mg | Main Study EFX 50 mg | Main Study EFX 70 mg | Main Study Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Percent change from baseline | -63.21 (5.01) | -70.92 (4.97) | -72.26 (5.04) | -0.29 (4.55)

4. Secondary Outcome: Main: Percent Change From Baseline in Hepatic Fat Fraction Measured by MRI-PDFF at Week 22-24.
Description: as for outcome 1
Time Frame: 22-24 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Main Study EFX 28 mg | Main Study EFX 50 mg | Main Study EFX 70 mg | Main Study Placebo
Number analyzed (Participants) | 16 | 17 | 15 | 2
Percent change from baseline | -49.80 (7.64) | -43.37 (7.52) | -63.70 (7.62) | -69.87 (20.78)

5. Secondary Outcome: Main: Responder: Subjects Who Achieved a Clinically Meaningful Relative Reduction of at Least 30% in Liver Fat Content as Measured by MRI-PDFF at Week 12.
Description: Main Study. The analyses included the treatment group and F1 fibrosis score (F1 vs F2-3) as factors and baseline hepatic fat fraction measured by MRI-PDFF as a covariate.
Time Frame: 12 weeks
Population: Full Analysis Set (all randomized subjects)
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study EFX 28 mg | Main Study EFX 50 mg | Main Study EFX 70 mg | Main Study Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
Participants | 16 | 17 | 15 | 2

6. Secondary Outcome: Main: Responder Based on NAFLD Activity Score System (NAS): Subjects Who Had a Decrease of ≥2 Points in NAS With at Least a 1-point Reduction in Either Lobular Inflammation or Hepatocellular Ballooning and With no Concurrent Worsening of Fibrosis Stage.
Description: Main study: Responders were defined for subjects with ≥ 30% relative fat reduction on MRI-PDFF at Week 12 and required to return between Weeks 22 - 24. Fisher's exact test was used for the analysis using the Full Analysis Set with missing values imputed as non-responders and repeated on Liver Biopsy Evaluable Analysis Set without imputation.
Time Frame: 22-24 weeks
Population: Liver Biopsy Evaluable Analysis Set (subjects from Full Analysis Set with Baseline and Week 22-24 liver biopsy results)
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study EFX 28 mg | Main Study EFX 50 mg | Main Study EFX 70 mg | Main Study Placebo
Number analyzed (Participants) | 13 | 13 | 14 | 2
Participants | 10 | 10 | 11 | 1

7. Secondary Outcome: Main: Change From Baseline in ALT at Week 12, 16, and 20.
Description: ANCOVA model with treatment group, baseline hepatic fat fraction (<15% vs ≥15%), and F1 fibrosis score (F1 vs F2-3) as factors and baseline value as a covariate.
Time Frame: 12, 16, and 20 weeks
Population: Full Analysis Set (all randomized subjects)
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Main Study EFX 28 mg | Main Study EFX 50 mg | Main Study EFX 70 mg | Main Study Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
U/L
  Change from Baseline to Week 12 | -24.46 (3.76) | -30.47 (3.59) | -32.29 (3.59) | -5.94 (3.38)
  Change from Baseline to Week 16 | -23.46 (4.87) | -31.99 (4.59) | -32.52 (4.65) | -3.17 (4.42)
  Change from Baseline to Week 20 | -17.57 (4.42) | -21.20 (4.17) | -28.70 (4.29) | -4.29 (3.96)

8. Secondary Outcome: Cohort C: Change From Baseline in Liver Stiffness as Evaluated by FibroScan at Week 16
Description: Cohort C: ANCOVA model with treatment group as a factor and baseline liver stiffness as evaluated by FibroScan® as a covariate using the Full Analysis Set. Missing values at Week 16 were imputed using the last-observed-carried-forward (LOCF) method.
Time Frame: 16 weeks
Population: Full Analysis Set (all randomized subjects)
Measure: Least Squares Mean (Standard Error); unit: KPa
Arm/Group | Cohort C EFX 50 mg | Cohort C Placebo
Number analyzed (Participants) | 20 | 10
KPa | -37.6 (8.6) | 12.1 (12.0)

9. Secondary Outcome: Cohort C: Change From Baseline in Non-invasive Biomarkers Including Pro-C3 at Week 12, 16, and 20.
Description: Cohort C. ANCOVA model with treatment group as a factor and baseline liver stiffness as evaluated by FibroScan® as a covariate using the Full Analysis Set. Missing values were imputed using the last-observed-carried-forward (LOCF) method.
Time Frame: 12, 16, and 20 weeks
Population: Full Analysis Set (all randomized subjects)
Measure: Least Squares Mean (Standard Error); unit: ug/L
Arm/Group | Cohort C EFX 50 mg | Cohort C Placebo
Number analyzed (Participants) | 20 | 10
ug/L
  Change from Baseline to Week 12 | -8.4 (1.1) | -2.8 (1.5)
  Change from Baseline to Week 16 | -9.0 (1.2) | -3.4 (1.7)
  Change from Baseline to Week 20 | -5.2 (1.2) | -4.9 (1.7)

10. Secondary Outcome: Cohort C: Change From Baseline in Non-invasive Biomarkers Including Liver Fibrosis by ELF Test Score at Week 12 and 16.
Description: Cohort C. The enhanced liver fibrosis (ELF) score describes the severity of liver fibrosis where a score of <7.7 indicates no or mild fibrosis, a score of ≥7.7 to <9.8 indicates moderate fibrosis, and a score of ≥9.8 indicates severe fibrosis. A change from baseline with a negative value indicates a decrease in severity of liver fibrosis.
  An ANCOVA model with treatment group as a factor and baseline liver stiffness as evaluated by FibroScan® as a covariate using the Full Analysis Set was used. Missing values were imputed using the last-observed-carried-forward (LOCF) method.
Time Frame: 12 and 16 weeks
Population: Full Analysis Set (all randomized subjects)
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Cohort C EFX 50 mg | Cohort C Placebo
Number analyzed (Participants) | 20 | 10
Score on a scale
  Change from Baseline to Week 12 | -0.3 (0.2) | 0.3 (0.2)
  Change from Baseline to Week 16 | -0.4 (0.1) | 0.3 (0.2)

ADVERSE EVENTS:
Time Frame: 20-24 weeks
Arm/Group | Main Study EFX 28 mg | Main Study EFX 50 mg | Main Study EFX 70 mg | Main Study Placebo | Cohort C EFX 50 mg | Cohort C Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/20 | 0/21 | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/19 | 1/20 | 0/21 | 0/20 | 1/10
Other Adverse Events (participants affected / at risk) | 18/19 | 17/19 | 19/20 | 16/21 | 19/20 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study EFX 28 mg (N=19) | Main Study EFX 50 mg (N=19) | Main Study EFX 70 mg (N=20) | Main Study Placebo (N=21) | Cohort C EFX 50 mg (N=20) | Cohort C Placebo (N=10)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study EFX 28 mg (N=19) | Main Study EFX 50 mg (N=19) | Main Study EFX 70 mg (N=20) | Main Study Placebo (N=21) | Cohort C EFX 50 mg (N=20) | Cohort C Placebo (N=10)
Diarrhea (Gastrointestinal disorders) | 5 | 11 | 7 | 4 | 10 | 1
Nausea (Gastrointestinal disorders) | 8 | 5 | 12 | 1 | 9 | 2
Vomiting (Gastrointestinal disorders) | 6 | 4 | 5 | 0 | 4 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 3 | 4 | 1 | 1 | 1
Frequent bowel movement (Gastrointestinal disorders) | 3 | 2 | 4 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 3 | 2
Constipation (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 4 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1 | 0
Feces soft (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 2
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Defecation Urgency (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Eosinophilic esophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 7 | 4 | 2 | 0
Injection site erythema (General disorders) | 2 | 1 | 5 | 0 | 5 | 0
Injection site reaction (General disorders) | 2 | 1 | 4 | 1 | 6 | 0
Injection site bruising (General disorders) | 2 | 1 | 1 | 1 | 4 | 1
Injection site pruritus (General disorders) | 2 | 0 | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 2 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Injection site irritation (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 2 | 0 | 0
Thirst (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Axillary pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Feeling of body temperature change (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Injection site hemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Edema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 2 | 3 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 3 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 0 | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 2 | 0 | 1 | 4 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Injection site cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Esophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 4 | 5 | 5 | 1 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 3 | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lack of satiety (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Food aversion (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 2 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 2 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin odor abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 3 | 3 | 4 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 1 | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hyperactive pharyngeal reflex (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 2 | 1 | 0 | 1 | 0
Weight increased (Investigations) | 1 | 1 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Occult blood positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Total lung capacity decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 1 | 0
Burns first degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Eyelid injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 3 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 3 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Retracted nipples (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eyelid edema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT03976401/Prot_000.pdf
  • Statistical Analysis Plan: Main Study (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT03976401/SAP_001.pdf
  • Statistical Analysis Plan: Cohort C (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT03976401/SAP_002.pdf